CLINICAL TRIAL: NCT06329440
Title: Comparison of Diaphragma Thickness and Perfusion Index Change in Supraclavicular and Costoclavicular Brachial Plexus Block in Adult Patients Undergoing Hand Surgery
Brief Title: Comparison of Supraclavicular and Costoclavicular Brachial Plexus Blocks in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, MD, Assoc Prof, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2023/880
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Diaphragm Injury
Keywords: regional anaesthesia; acute pain; peripheral block
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costoclavicular block (Active Comparator): Patients who will receive costoclavicular brachial plexus block for hand surgery. Costoclavicular block is performed via depositing local anesthetic in the costoclavicular space which is placed in the posterior of middle part of the clavicle. The diaphragma thickness will be evaluated after the surgery in postanesthesia care unit.
  Interventions: Diagnostic Test: Ultrasonographic measurement of diaphragm thickness
- Supraclavicular block (Active Comparator): Patients who will receive supraclavicular brachial plexus block for hand surgery. Supraclavicular is performed via depositing local anesthetic using corner pocket technique which is described as injecting the drugs to the inferolateral side of axillary artery above the 1st rib. The diaphragma thickness will be evaluated after the surgery in postanesthesia care unit.
  Interventions: Diagnostic Test: Ultrasonographic measurement of diaphragm thickness

INTERVENTIONS:
Diagnostic Test: Ultrasonographic measurement of diaphragm thickness — Lineer probe of the ultrasound machine will be placed sagitally on the level of 9th to 11th rib in order to observe diaphragmatic thickness change during a sniff. The thicknesses will be measured both in full expiration (Te) and full inspirium (Ti) in centimeters. The diaphragm thickness fraction will be calculated as follows: (Ti-Te)/Te

SUMMARY:
Hemidiaphragmatic paresis is a common side effect of brachial plexus blocks such as supraclavicular or infraclavicular block techniques. It has been shown that diaphragma thickness is affected at some extent in supraclavicular block and also in costoclavicular block which is accepted as an infraclavicular approach. However, these two approaches have not been extensively investigated before in terms of the diaphragmatic paresis. Here, it is aimed to compare these two methods considering their effects on diaphragma thickness in inspirium and in expirium. Moreover, the performance properties such as motor and sensory block onset, needle visualization time, needle visualization difficulty, postoperative pain scores, and lastly the perfusion index which is known to be reflecting vasodilation will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* adult patients who will undergone upper extremity peripheral block

Exclusion Criteria:

* coagulation disorders
* paediatric patients
* Patients who do not accept regional anaesthesia
* known local anaesthetic allergy
* Patients who are under anticoagulant therapy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Diaphragm thickness fraction (centimeters) | Up to 4 hours
  The formula is as follows: (Diaphragm thickness at the end of inspirium - Diaphragm thickness at the end of expirium)/ Diaphragm thickness at the end of expirium.
  This ratio gives the fraction of diaphragm thickness which reflects possible diaphragm paresis or paralysis. The thickness is measured during a sniff test via ultrasound for which the probe is placed sagitally on the level of 9th to 11th rib on the mid axillary line.

SECONDARY OUTCOMES:
Diaphragm thickness at the end of expirium (centimeters). | Up to 4 hours
  The thickness is measured during a sniff test via ultrasound for which the probe is placed sagitally on the level of 9th to 11th rib on the mid axillary line.
Diaphragm thickness at the end of inspirium (centimeters). | Up to 4 hours.
  The thickness is measured during a sniff test via ultrasound for which the probe is placed sagitally on the level of 9th to 11th rib on the mid axillary line.
Perfusion index change | Up to 4 hours
  Perfusion index is measured before and after peripheral block (10th, 20th, and 30th minute after block performance), and also at the end of the case. It is calculated as pulsatile signal (AC)X100/non-pulsatile signal (DC). This indicator shows the block related regional vasodilation. Both block techniques will be compared in this regard.
Motor and sensory block onset time | Up to 45 minute
  After performing the block, n.musculocutaneus, n.medianus, n.radialis, and n.ulnaris will be evaluated via physical examination every 5 minute.For the sensory evaluation, a blunt needle will be pinned on the relevant areas (median nerve: volar face of the middle finger, ulnar nerve: volar face of the 5th finger, radial nerve: hand dorsum and musculocutaneus nerve: lateral part of forearm), and scored as follows: 0: feels pain/absent sensorial blockade, 1: feels touch/partial blockade, 2: no sense/complete blockade. Motor activity will be evaluated via checking the motor response of the same branches and accordingly scoring was as follows: 0: no motor block, 1: partial motor block, 2: total motor block.
Postoperative pain scores (0-10) | Up to 24 hours
  Pain will be evaluated using numeric rating scale which is between 0 to 10 (0= no pain, 10=the worst pain experienced). This scale will be questioned in postoperative 1st, 2nd, 4th, 6th, 12th and 24th hours.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, MD, Assoc Prof, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided